CLINICAL TRIAL: NCT03073265
Title: Validation Study Protocol - Additional Study on Fresh Samples STA - Apixaban Calibrator & STA - Apixaban Control
Brief Title: Apixaban Validation Study - Additional Study on Fresh Samples
Status: Completed | Type: Observational
Sponsor: Diagnostica Stago (Industry)
Responsible Party: Sponsor
Other Study IDs: VSP A006 - US_comp / 1
Record Dates: First submitted 2017-02-27; First posted 2017-03-08 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2017-05

CONDITIONS: Anticoagulation With Apixaban
Keywords: DOAC; apixaban; IVD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients on apixaban: Patients currently on apixaban who meet inclusion/exclusion criteria A blood draw will be done on each patient to measure apixaban concentration in plasma using anti-Xa assay and LCMS.
  Interventions: Device: STA-Apixaban Calibrator & Control

INTERVENTIONS:
Device: STA-Apixaban Calibrator & Control — Measurement of apixaban level will be done using anti-Xa assay (IVD).

SUMMARY:
The objective is to demonstrate the performances of STA® - Apixaban Calibrator & STA® - Apixaban Control used in combination with STA® - Liquid Anti-Xa to measure apixaban concentration in plasma. Anti-Xa results will be compared to LCMS (liquid chromatography - mass spectrometry) for validation of the assay. For this study, the anti-Xa assay will be performed on fresh samples only.

The results will be used to complete results obtained previously on frozen samples.

DETAILED DESCRIPTION:
About 60 samples from patients on apixaban meeting inclusion/exclusion criteria will be included in this study. Two sites will be in charge of sample recruitment and anti-Xa testing. A third site will be in charge of LCMS testing.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years,
* Weight ≤ 60 kg,
* Haematocrit below normal values as determined by local laboratory or < 40% for male and < 37% for female
* Renal impairment documented (creatinine clearance ≤ 80 mL/min as per Cockcroft -Gault equation) or serum creatinine ≥ 1.5 mg/dL
* Co-medication with aspirin or any other NSAIDs (nonsteroidal anti-inflammatory drugs)
* Co-medication with anti-platelet agents

Exclusion Criteria:

* Patients less than 18 years old
* Patients under other anti-coagulant treatment
* Samples that are not collected, stored, or handled in accordance with sample collection procedures defined above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with apixaban presenting at least one of the listed inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Method comparison between Anti-Xa method and LCMS to measure apixaban in plasma | The anti-Xa assay will be tested within 6h after sample collection and LCMS will be performed on frozen samples, at maximum 2 months after collection.
  Compare results from anti-Xa assay and LCMS to measure apixaban in plasma samples. Regression and difference charts will be used to compare the methods.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Moses Cone Memorial Hospital, Greensboro, North Carolina
  - Lehigh Valley Health Nrwork, Allentown, Pennsylvania